CLINICAL TRIAL: NCT00915824
Title: Prevention of Potentially Inappropriate Prescribing in Late Life Using STOPP (Screening Tool of Older Persons' Potentially Inappropriate Prescriptions) and START (Screening Tool to Alert Doctors to Right i.e. Appropriate Indicated Treatment): A Randomized Controlled Trial.
Brief Title: Prevention of Potentially Inappropriate Prescribing in Late Life Using Screening Tool of Older Persons' Potentially Inappropriate Prescriptions (STOPP) and Screening Tool to Alert Doctors to Right Treatment (START) Criteria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cork University Hospital (Other)
Responsible Party: Dr. Paul Gallagher, Clinical Research Fellow, Department of Geriatric Medicine, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CRT2006029
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: Drug therapy; Prescribing; Appropriateness; Randomized controlled trial; STOPP/START criteria; Appropriateness of prescribing in older patients; Prescription Drugs
MeSH Terms: interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STOPP/START intervention (Experimental): STOPP/START intervention group
  Interventions: Other: STOPP/START criteria

INTERVENTIONS:
Other: STOPP/START criteria — Application of STOPP/START criteria to the patient's prescription and diagnostic information with subsequent written recommendation on pharmaceutical care to the patient's medical team

SUMMARY:
Potentially inappropriate prescribing is common in older patients and encompasses overuse, misuse and underuse of medications. Potentially inappropriate prescribing is associated with negative outcomes including adverse drug events and hospitalization.

STOPP (Screening Tool of Older Person's potentially inappropriate Prescriptions) and START (Screening Tool to Alert doctors to Right Treatment) is a new screening tool designed to detect instances of potentially inappropriate medication use and under-prescribing of clinically indicated medications in older patients. The purpose of this study is to determine whether clinical implementation of STOPP/START criteria in hospitalized older patients is effective in improving prescribing quality.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 65 years and older admitted to the general medical services of Cork University Hospital, Cork, Ireland

Exclusion Criteria:

* Patient admitted to a geriatric medicine service, psychiatry of old age service or clinical pharmacology service, or under review of these services during the previous 12 months
* Critically ill patient (admitted to the intensive care unit)
* Terminally ill patient
* Refusal of patient or hospital physician to participate
* No time for the research physician to enrol the patient within 3 days of admission

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Appropriateness of prescribing using the Medication Appropriateness Index and the Assessment of Underutilization of Medication Tool | Measured on admission, discharge and at 2, 4 and 6 months post-discharge

SECONDARY OUTCOMES:
Composite health resource utilization including hospital readmission and primary care consultations | at 2, 4 and 6 months post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gallagher, MB MRCPI, Principal Investigator — Cork University Hospital; Denis O'Mahony, MD FRCPI, Study Director — Cork University Hospital
Locations (1):
- Cork University Hospital, Cork, Ireland